CLINICAL TRIAL: NCT00753571
Title: Cistanche Total Glycosides Treatment for Amyotrophic Lateral Sclerosis: A Randomized Control Trial Study Assessing Clinical Response
Brief Title: Cistanche Total Glycosides for Amyotrophic Lateral Sclerosis: A Randomized Control Trial (RCT) Study Assessing Clinical Response
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Dongsheng Fan, MD, Peiking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PUTH-1
Record Dates: First submitted 2008-09-15; First posted 2008-09-16 (Estimated); Last update posted 2009-12-30 (Estimated); Status verified 2008-09

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; Cistanche Total Glycosides; Randomized Control Trial Study
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 1,CTG,po
  Interventions: Drug: Cistanche Total Glycosides
- 2 (Placebo Comparator)
  Interventions: Drug: Cistanche Total Glycosides

INTERVENTIONS:
Drug: Cistanche Total Glycosides — Drug: Cistanche Total Glycosides Cistanche Total Glycosides ,1.8g/day(6 capsules) po Qd*9months Arms: 1 Drug: blank capsules 6 capsules po Qd*9months
  Arms: 2

SUMMARY:
This study will examine the effectiveness of Cistanche Total Glycosides(CTG) in treating patients with amyotrophic lateral sclerosis (ALS) - a fatal neurological degenerative disease that causes adult-onset, progressive motor neurons loss in the spinal cord, brain stem and motor cortex. Patients develop progressive wasting and weakness of both upper and lower limbs, bulbar and respiratory muscles. Usually death from respiratory failure typically is within 3-5 years of diagnosis. Although there are various treatments for ALS, riluzole is the only approved treatment to delay the disease progression. Cistanche Total Glycosides is an approved drug that has protective effects. It acts anti-apoptosis by activating several protective pathways, stimulates neuronal differentiation of adult neural stem cells in the brain, and improves long-term recovery. CTG is a highly attractive candidate for the treatment of neurodegenerative conditions such as ALS.

Patients 18 to 65 years of age who have had mild to moderately severe ALS for 0.5 to 2 years of duration may be eligible for this study. Candidates will be screened with a medical history and possible review of medical records, physical examination, blood test, urine and stool analyses, electrocardiogram, electrophysiological examination, neurological imaging and, for women, a pregnancy test.

Participants will have drug therapy according to randomized number. One group receives CTG while other group receives placebo. For the procedure, patients are given a medication to lessen anxiety and any discomfort. Patients receive drugs for 9 months. The CTG dosage is 1.8g/day. Physical examination and interview, Appel ALS scale and ALS-Functional Rating Scale will be done in 28 days and 3, 6, 9months. Electrophysiological examination will be tested per 3 months. Blood samples will be collected on treat28 days and 3, 6, 9months.

DETAILED DESCRIPTION:
This study will examine the effectiveness of Cistanche Total Glycosides(CTG) in treating patients with amyotrophic lateral sclerosis (ALS) - a fatal neurological degenerative disease that causes adult-onset, progressive motor neurons loss in the spinal cord, brain stem and motor cortex. Patients develop progressive wasting and weakness of both upper and lower limbs, bulbar and respiratory muscles. Usually death from respiratory failure typically is within 3-5 years of diagnosis. Although there are various treatments for ALS, riluzole is the only approved treatment to delay the disease progression. Cistanche Total Glycosides is an approved drug that has protective effects. It acts anti-apoptosis by activating several protective pathways, stimulates neuronal differentiation of adult neural stem cells in the brain, and improves long-term recovery. CTG is a highly attractive candidate for the treatment of neurodegenerative conditions such as ALS.

Patients 18 to 65 years of age who have had mild to moderately severe ALS for 0.5 to 2 years of duration may be eligible for this study. Candidates will be screened with a medical history and possible review of medical records, physical examination, blood test, urine and stool analyses, electrocardiogram, electrophysiological examination, neurological imaging and, for women, a pregnancy test.

Participants will have drug therapy according to randomized number. One group receives CTG while other group receives placebo. For the procedure, patients are given a medication to lessen anxiety and any discomfort. Patients receive drugs for 9 months. The CTG dosage is 1.8g/day. Physical examination and interview, Appel ALS scale and ALS-Functional Rating Scale will be done in 28 days and 3, 6, 9months. Electrophysiological examination will be tested per 3 months. Blood samples will be collected on treat28 days and 3, 6, 9months.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must have a verifiable diagnosis of ALS of 0.5 to 2 years' duration.
* The diagnosis must be supported by the Revised Criteria of the World Federation of Neurology.
* The grades of diagnosis must be clinically definite ALS or clinically probable ALS.
* All subjects must be over age 18 and below 65.
* The ALS is mildly to moderate based on ALS Health State Scale.
* Electrophysiological features show CMAP amplitude of motor nerve normal or mild declining.
* Serum creatine kinase is normal or mild upper, less than 500U/L.

Exclusion Criteria:

* If anyone of the above eligibility requirements is not met
* Use of any other investigational agent within 30 days beginning the treatment phase of this study
* Severe cardiac, pulmonary, hepatic or/and hematic disease
* HIV positivity or signs and symptoms consistent with HIV infection
* Pregnant or nursing women
* History of cancer with less than 5 years documentation of a disease-free state
* History of anaphylactic reaction or hypersensitivity to G-CSF or proteins derived from E.coli
* Alcohol or drug abuse in recent 1 year
* Can't understand or obey the rules of treatment
* Blood donor in recent 30 days

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-12 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
The mean rate of decline of ALS-FRS score | 12 months

SECONDARY OUTCOMES:
The mean rate decline of the AARS score | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Dongsheng Fan, MD; Liping Wang,MD, Beijing, Beijing Municipality, China

REFERENCES:
- See also: Related Info — http://www.als.net/